CLINICAL TRIAL: NCT04377269
Title: Short-Term and Long-Term Effects of Ankle Joint Taping and Bandaging on Balance, Proprioception and Vertical Jump Among Volleyball Players With Chronic Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Gelisim University (Other)
Responsible Party: Principal Investigator, Motaz Alawna, Assistant Professor (Principal Investigator), Istanbul Gelisim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Taping, Bandaging, Volleyball
Record Dates: First submitted 2020-05-02; First posted 2020-05-06 (Actual); Last update posted 2020-05-07 (Actual); Status verified 2020-05

CONDITIONS: Chronic Ankle Instability

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Taping Group (Experimental): 33 participants, received ankle taping
  Interventions: Other: Taping and Bandaging
- Bandaging (Experimental): 33 participants, received ankle bandaging
  Interventions: Other: Taping and Bandaging
- Placebo Taping (Control) Group (Placebo Comparator): 34 participants, received ankle placebo taping
  Interventions: Other: Taping and Bandaging

INTERVENTIONS:
Other: Taping and Bandaging — Ankle taping: a hard preventive Zinc oxide tape was used. The taping procedures consisted of three separate steps. 1) included the application of the anchor tape. 2) application of the stirrup tape. The stirrup tape was performed two times by holding the foot in a neutral position and the tape is placed as it passed through the medial side of the ankle (under the foot), just over the heel area (posterior one-third of the foot) and up along the lateral side of the ankle. Bandaging: standard 10cm width elastic bandage used. The bandage wrapped around the ankle joint in the form of an 8-figure. Bandage started from the forefoot, moving diagonally upwards and steeply enough to go well above the heel to end around the lower calf area to form an anchor. Then, it moved diagonally down across the mid-foot. Placebo: 10cm long tape was applied on the lateral side of the leg, just above the lateral malleolus and aligned with peroneus longus tendon

SUMMARY:
Objective: This study aimed to 1) investigate the long-term effect of taping and bandaging on proprioception, balance, and vertical jump among volleyball players with ankle instability, 2) Compare the short-term effects of taping and bandaging on these outcome measures, 3) Compare the long-term effects of taping and bandaging on these outcome measures.

Design: A single-blinded randomized controlled study Setting: Rehabilitation Laboratory at Istanbul Gelisim University, Turkey Subjects: One-hundred participants with a chronic ankle sprain (CAI) Primary outcome measures: Proprioception (ankle range of motion absolute error), balance(Y-balance test), and vertical jump (vertical jump tester) Interventions: Participants were distributed into three groups: taping group (n=33) received ankle rigid taping, bandaging group (n=33) received ankle bandaging, and control group (n=34) received placebo taping. All three previous external supports were applied for 8 weeks. The measurements were performed at baseline, immediately after applying for support, two weeks after support and eight months after support.

ELIGIBILITY:
Inclusion Criteria:

* Volleyball Player
* 18-30 years old
* Athletes with chronic ankle instability

Exclusion Criteria:

* Previous hip/pelvis knee, or foot surgery within the past year
* Leg length discrepancies
* Known balance impairment due to neurological disorder
* Vestibular disorder
* Pregnancy
* Brain concussion within the previous three months
* Taking any medication that may affect alertness or balance

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Proprioception | 2 Months
  Measure the Range of motion Standard error at three different range of motion angles (10° dorsiflexion, neutral position, 10° plantarflexion, and 20° plantarflexion).
Balance | 2 Months
  The Y-Balance test was used to evaluate balance.
Vertical Jump Distance | 2 Months
  The vertical jump tester (Sports Imports, Columbus, OH)

IPD SHARING:
Plan to Share IPD: No